CLINICAL TRIAL: NCT02055183
Title: Botulinum Antitoxin Patient Registry for the Evaluation of Safety and Clinical Outcomes of Pediatric and Adult Patients Following BAT Treatment for Confirmed or Suspected Exposure to Botulinum Toxin.
Brief Title: BT-010 Registry for the Evaluation of Safety and Clinical Outcomes in Patients Treated With Botulinum Antitoxin
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: BT-010
Record Dates: First submitted 2014-01-29; First posted 2014-02-05 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Botulism
Keywords: Registry; Botulinum antitoxin; Botulism Antitoxin Heptavalent- (Equine); BAT®
MeSH Terms: conditions — Botulism | interventions — Botulinum Antitoxin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with BAT®: Any patient of any age with a confirmed or suspected exposure to botulinum toxin who were treated with BAT®.
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: BAT — Noninterventional, retrospective, observational phase 4 patient Registry
  Other Names: Botulism Antitoxin

SUMMARY:
The purpose of the Registry was to evaluate patient safety following Botulism Antitoxin Heptavalent (A, B, C, D, E, F, G) - (Equine) (BAT®) administration in adult and pediatric patients with a confirmed or suspected exposure to botulinum toxin.

DETAILED DESCRIPTION:
A full description of the patient registry can be found in the paper titled: Safety and Clinical Outcomes of an Equine-derived Heptavalent Botulinum Antitoxin Treatment for Confirmed or Suspected Botulism in the United States. Richardson JS, Parrera GS, Astacio H, Sahota H, Anderson DM, Hall C, Babinchak T. Clin Infect Dis. 2019 Apr 15;70(9):1950-1957.

ELIGIBILITY:
Inclusion Criteria:

* Any patient of any age [age category: pediatric-newborn infants (0 to 27 days), infants and toddlers (28 days to 23 months), children (2 to 11-years), and adolescents (12 to <17-years); adult (17-64-years); and geriatric (≥65-years)] with a confirmed or suspected exposure to botulinum toxin who were treated with BAT® provided by the CDC.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient of any age [age category: pediatric-newborn infants (0 to 27 days), infants and toddlers (28 days to 23 months), children (2 to 11-years), and adolescents (12 to <17-years); adult (17-64-years); and geriatric (≥65-years)] with a confirmed or suspected exposure to botulinum toxin who were treated with BAT® provided by the CDC.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious adverse events | From BAT® administration up to discharge from hospital (200 days)
  The data obtained will more clearly define the absolute risk (incidence rates) of hypersensitivity/allergic reactions, including serum sickness, febrile reactions, hemodynamic instability, bradycardia, and other serious adverse events in pediatric and adult patients that are treated with BAT® due to a confirmed or suspected case of botulism.

OTHER OUTCOMES:
Number of participants developing acute hypersensitivity | 24 hours
  Reactions that may occur shortly after exposure to BAT® and can include, but are not limited to, urticaria, pruritus, erythema, angioedema, bronchospasm with wheezing or cough, stridor, laryngeal edema, hypotension, or tachycardia.
Number of participants developing anaphylaxis /anaphylactoid reactions | 24 hours
  Severe form of acute, severe hypersensitivity reaction with multiorgan system involvement that occurs with sudden onset after exposure to an allergen. Case definition of anaphylaxis requires a sudden onset and rapid progression of signs and symptoms and involvement of multiple (≥ 2) organ systems (cardiovascular, dermatological or respiratory).
Number of participants developing delayed allergic reaction or serum sickness | 10-21 days
  This includes symptoms such as, but not limited to, fever, urticarial or maculopapular rash, myalgia, arthralgia, and lymphadenopathy occurring 10-21 days after BAT® infusion.
Number of participants developing infusion reactions | 24 hours
  Infusion reactions are unexpected reactions that cannot be explained by the known toxicity profile of the drug. Infusion reactions are the result of the infusion process (rate, volume, etc.) and are often referred to as "hypersensitivity reactions" as well. In the absence of an allergic component, the term "infusion reaction" is preferred. Infusion reactions may affect any organ system in the body. Most are mild in severity, although severe and fatal reactions may occur. The most common signs and symptoms may include, but are not limited to flushing, itching, alterations in heart rate and blood pressure, dyspnea or chest discomfort, back or abdominal pain, fever and/or shaking chills (rigors), nausea, vomiting, and/or diarrhea, skin rashes, throat tightening, hypoxia, seizures, dizziness and/or syncope.
Number of participants developing febrile reactions | 1 hour
  Febrile reaction is an absolute temperature > 38.1°C or an increase in temperature >1°C above baseline temperature that occurs during or within 1 hour of BAT® infusion and is unrelated to the underlying illness.
Number of participants developing hemodynamic instability | 24 hours
  A state requiring pharmacologic or mechanical support to maintain a normal blood pressure or adequate cardiac output.
Number of participants developing bradycardia | 24 hours
  Bradycardia is defined as an abnormally slow heart rate; usually <60 beats per minute in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Richardson, Ph.D., Study Chair — Emergent BioSolutions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnon SS, Schechter R, Inglesby TV, Henderson DA, Bartlett JG, Ascher MS, Eitzen E, Fine AD, Hauer J, Layton M, Lillibridge S, Osterholm MT, O'Toole T, Parker G, Perl TM, Russell PK, Swerdlow DL, Tonat K; Working Group on Civilian Biodefense. Botulinum toxin as a biological weapon: medical and public health management. JAMA. 2001 Feb 28;285(8):1059-70. doi: 10.1001/jama.285.8.1059. PMID 11209178
- [Background] Black RE, Gunn RA. Hypersensitivity reactions associated with botulinal antitoxin. Am J Med. 1980 Oct;69(4):567-70. doi: 10.1016/0002-9343(80)90469-6. PMID 7191633
- [Background] Gangarosa EJ, Donadio JA, Armstrong RW, Meyer KF, Brachman PS, Dowell VR. Botulism in the United States, 1899-1969. Am J Epidemiol. 1971 Feb;93(2):93-101. doi: 10.1093/oxfordjournals.aje.a121239. No abstract available. PMID 4925448
- [Background] Lack JA, Stuart-Taylor ME. Calculation of drug dosage and body surface area of children. Br J Anaesth. 1997 May;78(5):601-5. doi: 10.1093/bja/78.5.601. PMID 9175982
- [Background] Lieberman P, Nicklas RA, Oppenheimer J, Kemp SF, Lang DM, Bernstein DI, Bernstein JA, Burks AW, Feldweg AM, Fink JN, Greenberger PA, Golden DB, James JM, Kemp SF, Ledford DK, Lieberman P, Sheffer AL, Bernstein DI, Blessing-Moore J, Cox L, Khan DA, Lang D, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph C, Schuller DE, Spector SL, Tilles S, Wallace D. The diagnosis and management of anaphylaxis practice parameter: 2010 update. J Allergy Clin Immunol. 2010 Sep;126(3):477-80.e1-42. doi: 10.1016/j.jaci.2010.06.022. Epub 2010 Aug 7. PMID 20692689
- [Background] Ruggeberg JU, Gold MS, Bayas JM, Blum MD, Bonhoeffer J, Friedlander S, de Souza Brito G, Heininger U, Imoukhuede B, Khamesipour A, Erlewyn-Lajeunesse M, Martin S, Makela M, Nell P, Pool V, Simpson N; Brighton Collaboration Anaphylaxis Working Group. Anaphylaxis: case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5675-84. doi: 10.1016/j.vaccine.2007.02.064. Epub 2007 Mar 12. No abstract available. PMID 17448577
- [Background] Schleis TG. Interference of maltose, icodextrin, galactose, or xylose with some blood glucose monitoring systems. Pharmacotherapy. 2007 Sep;27(9):1313-21. doi: 10.1592/phco.27.9.1313. PMID 17723085
- [Background] Shapiro RL, Hatheway C, Swerdlow DL. Botulism in the United States: a clinical and epidemiologic review. Ann Intern Med. 1998 Aug 1;129(3):221-8. doi: 10.7326/0003-4819-129-3-199808010-00011. PMID 9696731
- [Background] Tacket CO, Shandera WX, Mann JM, Hargrett NT, Blake PA. Equine antitoxin use and other factors that predict outcome in type A foodborne botulism. Am J Med. 1984 May;76(5):794-8. doi: 10.1016/0002-9343(84)90988-4. PMID 6720725
- [Result] Richardson JS, Parrera GS, Astacio H, Sahota H, Anderson DM, Hall C, Babinchak T. Safety and Clinical Outcomes of an Equine-derived Heptavalent Botulinum Antitoxin Treatment for Confirmed or Suspected Botulism in the United States. Clin Infect Dis. 2020 Apr 15;70(9):1950-1957. doi: 10.1093/cid/ciz515. PMID 31209461
- See also: Morbidity and Mortality Weekly Report Center for Disease Control and Prevention. Investigational heptavalent botulinum antitoxin (HBAT™) to replace licensed botulinum antitoxin AB and investigational botulinum antitoxin E. — http://www.cdc.gov/mmwr/pdf/wk/mm5910.pdf
- See also: Botulism Antitoxin Heptavalent (A, B, C, D, E, F, G) - (Equine) (BAT™) United States Prescribing Information, 03/2013. — http://www.fda.gov/downloads/BiologicsBloodVaccines/BloodBloodProducts/ApprovedProducts/LicensedProductsBLAs/FractionatedPlasmaProducts/UCM345147.pdf